CLINICAL TRIAL: NCT04819438
Title: Comparative Bioavailability Study of a New Riluzole Orodispersible Film vs. a Marketed Oral Reference (Rilutek® Tablets) in Healthy Male and Female Volunteers
Brief Title: Riluzole Orodispersible Film Replicate Bioavailability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cross Research S.A. (Industry)
Collaborators: Zambon SpA (Industry)
Responsible Party: Principal Investigator, Milko Radicioni, Principal Investigator, Cross Research S.A.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Z7251J01
Record Dates: First submitted 2021-03-08; First posted 2021-03-29 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants
Keywords: Bioequivalence; Riluzole; Orodispersible film
MeSH Terms: interventions — Riluzole

STUDY DESIGN:
Intervention Model Description: The study was designed in agreement with the EMA guideline "Guidance on the investigation of bioequivalence", CPMP/EWP/QWP/1401/98 Rev. 1 January 2010 (9).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference/Test/Reference/Test (Experimental): Riluzole orodispersible film (test): The subjects will be treated with one orodispersible film containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence Rilutek® (reference): The subjects will be treated with one film-coated tablet containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence.
  Interventions: Drug: Riluzole 50 mg orodispersible film; Drug: Rilutek® 50 mg riluzole tablets
- Test/Reference/Test/Reference (Experimental): Riluzole orodispersible film (test): The subjects will be treated with one orodispersible film containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence Rilutek® (reference): The subjects will be treated with one film-coated tablet containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence.
  Interventions: Drug: Riluzole 50 mg orodispersible film; Drug: Rilutek® 50 mg riluzole tablets

INTERVENTIONS:
Drug: Riluzole 50 mg orodispersible film — Before each administration, the subjects will drink 20 mL of still mineral water in order to wet their mouth. Afterwards, using gloves, the investigator or deputy will take the orodispersible film (32.0x22.0 mm) out of the provided pouch and place the product directly on the top surface (dorsal aspect) of the subjects' tongue.
  Other Names: Test product (T)
Drug: Rilutek® 50 mg riluzole tablets — One film-coated tablet will be swallowed (without chewing) with 150 mL of still mineral water.
  Other Names: Reference product (R)

SUMMARY:
The objective of the study is to compare the pharmacokinetic profile of riluzole after replicate single dose of the novel orodispersible film test formulation and of the marketed reference Rilutek® tablets and to evaluate their bioequivalence.

DETAILED DESCRIPTION:
The new formulation riluzole orodispersible film is expected to fill an important medical need, since the medication can be easily administered without water and may improve patient care. Riluzole orodispersible film is easily administered, because the patient or caregiver needs only to place the film on the tongue, where it can immediately dissolve into the saliva and be ingested with intentional swallowing or during the normal reflex of swallowing, thus eliminating the need for swallowing a tablet with liquid or crushing it into soft food.

Zambon S.p.A., Italy, is sponsoring the present bioequivalence study in order to investigate the bioequivalence of the novel unit-dose product versus Rilutek® tablets, commercially available in Europe as 50 mg tablets. The dose strength for the test formulation is 50 mg, matching the 50 mg strength of the reference formulation.

The subjects will receive single oral doses of 50 mg of riluzole, as test orodispersible film and reference film-coated tablets, under fasting conditions, in each of 4 subsequent periods separated by wash-out intervals of at least 7 days between consecutive administrations, according to a 2-treatment, 4-period, replicate cross-over design.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the study
2. Sex and Age: men/women, 18-55 years old inclusive
3. Tobacco: non-smokers for at least 6 months prior to study screening
4. Body Mass Index (BMI): 18.5-29 kg/m2 inclusive
5. Vital signs: systolic blood pressure (SBP) 100-139 mmHg, diastolic blood pressure (DBP) 50-89 mmHg, heart rate 50-90 bpm, measured after 5 min at rest in the sitting position
6. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
7. Contraception and fertility (women only): women of child-bearing potential must be using at least one of the following reliable methods of contraception:

   1. A non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit
   2. A male sexual partner who agrees to use a male condom with spermicide
   3. A sterile sexual partner Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted. For all women, pregnancy test result must be negative at screening.

Exclusion Criteria:

1. Electrocardiogram (ECG) 12-leads: (supine position) clinically significant abnormalities; corrected QT interval > 450 msec
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
3. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness
4. Cotinine: positive cotinine test at screening
5. Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers may affect the outcome of the study
6. Diseases: clinically significant history or presence of renal, hepatic, gastrointestinal, cardiovascular, cerebrovascular, immunological, musculoskeletal, respiratory, skin, haematological, endocrine, psychiatric or neurological diseases or surgeries that may interfere with the aim of the study. Gastrointestinal pathologies include any clinically significant disorder of the mouth, e.g. impairment of swallowing, lesions, ulcerations, deformities, untreated dental caries
7. Dentures: presence of mouth jewellery, dentures, braces, piercings that may interfere with successful completion of the dosing
8. Medications: medications, including over the counter medications and herbal remedies for 2 weeks before study screening; central nervous system depressants, including opioids, benzodiazepines, general anaesthetics and anticonvulsants, or cytochrome C inhibitors, including cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, ketoconazole, diltiazem and antiretroviral agents, or strong cytochrome C inducers, including barbiturates, carbamazepine, glucocorticoids, phenytoin, St John's wort and rifampin, or hormonal oral or transdermal contraceptives for 30 days before study screening; implanted, injected, intravaginal or intrauterine hormonal contraceptives for 6 months before study screening
9. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
10. Blood donation: blood donations for 3 months before this study
11. Drug, alcohol, caffeine, tobacco: history of drug, alcohol [>1 drink/day for females and >2 drinks/day for males, defined according to the Dietary Guidelines 2015 ], caffeine (>5 cups coffee/tea/day) or tobacco use including any tobacco product like e-cigarettes and vamping products
12. Drug test: positive result at the drug test at screening or Day -1
13. Alcohol test: positive alcohol breath test at Day -1
14. Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians and vegans
15. Pregnancy (women only): positive or missing pregnancy test at screening or Day -1, pregnant or lactating women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-03-14 (Actual); Study Completion 2021-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — CROSS Research SA
Locations (1):
- CROSS Research SA Phase 1 Unit, Arzo, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the Phase I Unit from January 2021 to February 2021.
Pre-assignment Details: Fifty-four (54) subjects were randomised in the study and 53 of them received at least one dose of investigational product, while one subject discontinued the study before receiving any treatment due to adverse event.
Groups:
- Riluzole 50mg (Test) / Rilutek 50mg (Reference) / Riluzole 50mg (Test) / Rilutek 50mg (Reference): Riluzole 50 mg Orodispersible Film (Test, T): The subjects were treated with one orodispersible film containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence. Before each administration, the subjects drank 20 mL of still mineral water in order to wet their mouth. Afterwards, using gloves, the investigator or deputy took the orodispersible film (32.0x22.0 mm) out of the provided pouch and placed the product directly on the top surface (dorsal aspect) of the subjects' tongue.
  Rilutek 50 mg Tablet (Reference, R): The subjects were treated with one film-coated table containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence. One film-coated tablet was swallowed (without chewing) with 150 mL of still mineral water.
- Rilutek 50mg (Reference) / Riluzole 50mg (Test) / Rilutek 50mg (Reference) / Riluzole 50mg (Test): Riluzole 50 mg Orodispersible Film (Test, T): The subjects were treated with one orodispersible film containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence. Before each administration, the subjects drank 20 mL of still mineral water in order to wet their mouth. Afterwards, using gloves, the investigator or deputy took the orodispersible film (32.0x22.0 mm) out of the provided pouch and placed the product directly on the top surface (dorsal aspect) of the subjects' tongue.
  Rilutek 50 mg Tablet (Reference, R): The subjects were treated with one film-coated tablet containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence. One film-coated tablet was swallowed (without chewing) with 150 mL of still mineral water.
Period: Overall Study
Arm/Group | Riluzole 50mg (Test) / Rilutek 50mg (Reference) / Riluzole 50mg (Test) / Rilutek 50mg (Reference) | Rilutek 50mg (Reference) / Riluzole 50mg (Test) / Rilutek 50mg (Reference) / Riluzole 50mg (Test)
Started | 27 | 27
Completed | 26 | 25
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: The subjects will be treated with one orodispersible film containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence.
  The subjects will be treated with one film-coated table containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence.
  The subjects received single oral doses of 50 mg of riluzole, as test orodispersible film and reference film-coated tablets under fasting conditions, in each of 4 subsequent periods separated by wash-out intervals of at least 7 days between consecutive administrations, according to a 2-treatment, 4-period, replicate cross-over design.
Arm/Group | All Study Participants
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 51
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 54
Body weight [Mean (Standard Deviation); unit: kilograms] | 65.86 (10.87)
Height [Mean (Standard Deviation); unit: centimeters] | 167.8 (8.9)
Body mass index [Mean (Standard Deviation); unit: kilograms/square meters] | 23.30 (2.65)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Bioequivalent Rate of Absorption (Cmax) of Riluzole After Replicate Single Dose Administration of Test and Reference
Description: For each individual, the maximum plasma concentration (Cmax) of riluzole after replicate single dose administration of Test and Reference was measured. The Cmax 90% confidence interval of the ratio Test/Reference of the population means was calculated. The bioequivalence is demonstrated when the 90% confidence Interval of this ratio lies within the range 80.00-125.00% (acceptance interval).
Time Frame: 0 h (pre-dose) and 15, 30, 45 min, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24 and 36 h after the drug administration
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Riluzole Orodispersible Film (Test): The subjects will be treated with one orodispersible film containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence.
- Rilutek® Tablet (Reference): The subjects will be treated with one film-coated table containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence.
Arm/Group | Riluzole Orodispersible Film (Test) | Rilutek® Tablet (Reference)
Number analyzed (Participants) | 51 | 51
ng/mL | 315.62 (124.95) | 278.81 (123.32)
Statistical Analysis 1: Comparison: Riluzole Orodispersible Film (Test) vs Rilutek® Tablet (Reference); Test type: Equivalence — Acceptance criterion for bioequivalence analysis was that the 90% confidence interval for the Test/Reference ratio of Cmax geometric means was within the 80.00-125.00 range; p < 0.0001, ANOVA; Geometric Mean Ratio = 117.05, 90% CI 2-sided [110.43 to 124.06]

2. Primary Outcome: Evaluation of the Bioequivalent Extent of Absorption (AUC0-t) of Riluzole After Replicate Single Dose Administration of Test and Reference.
Description: For each individual, the area under the concentration-time curve from single dose Test and Reference administration to the last observed concentration time t (AUC0-t) of riluzole was measured. The AUC0-t 90% confidence interval of the ratio Test/Reference of the population means was calculated. The bioequivalence is demonstrated when the 90% confidence Interval of this ratio lies within the range 80.00-125.00% (acceptance interval).
Time Frame: 0 h (pre-dose), 15, 30, 45 min, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24 and 36 h after drug administration
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Riluzole Orodispersible Film (Test) | Rilutek® Tablet (Reference)
Number analyzed (Participants) | 51 | 51
h*ng/mL | 1263.40 (571.58) | 1135.98 (514.98)
Statistical Analysis 1: Comparison: Riluzole Orodispersible Film (Test) vs Rilutek® Tablet (Reference); Test type: Equivalence — Acceptance criterion for bioequivalence analysis was that the 90% confidence interval for the Test/Reference ratio of AUC0-t geometric means was within the 80.00-125.00 range; p < 0.0001, ANOVA; Geometric Mean Ratio = 111.82, 90% CI 2-sided [108.25 to 115.50]

3. Secondary Outcome: To Describe the t1/2 (Half-life) of Riluzole After Replicate Single Dose Administration of Test and Reference
Description: To Describe the half-life of riluzole, calculated, if feasible, as ln2/λz, After Replicate Single Dose Administration of Test and Reference.
Time Frame: 0 h (pre-dose), 15, 30, 45 min, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24 and 36 h after drug administration
Measure: Mean (Standard Deviation); unit: h
Groups:
- Riluzole Orodispersible Film (Test): The subjects were treated with one orodispersible film containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence
  Riluzole 50 mg Oral Film: Before each administration, the subjects drank 20 mL of still mineral water in order to wet their mouth. Afterwards, using gloves, the investigator or deputy took the orodispersible film (32.0x22.0 mm) out of the provided pouch and placed the product directly on the top surface (dorsal aspect) of the subjects' tongue.
- Rilutek® Tablet (Reference): The subjects were treated with one film-coated table containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence
  Rilutek 50Mg Tablet: One film-coated tablet was swallowed (without chewing) with 150 mL of still mineral water.
Arm/Group | Riluzole Orodispersible Film (Test) | Rilutek® Tablet (Reference)
Number analyzed (Participants) | 51 | 51
h | 10.22 (1.66) | 10.22 (1.48)

4. Secondary Outcome: To Describe the AUC0-∞ of Riluzole After Replicate Single Dose Administration of Test and Reference
Description: For each individual, the area under the concentration-time curve extrapolated to infinity after single dose administration of Test and Reference (AUC0-∞) was measured. The AUC0-∞ 90% confidence interval of the ratio Test/Reference of the population means was calculated. The bioequivalence is demonstrated when the 90% confidence Interval of this ratio lies within the range 80.00-125.00% (acceptance interval).
Time Frame: 0 h (pre-dose), 15, 30, 45 min, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24 and 36 h after drug administration
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Riluzole Orodispersible Film (Test) | Rilutek® Tablet (Reference)
Number analyzed (Participants) | 51 | 51
h*ng/mL | 1348.31 (630.80) | 1207.79 (566.13)
Statistical Analysis 1: Comparison: Riluzole Orodispersible Film (Test) vs Rilutek® Tablet (Reference); Test type: Equivalence — Acceptance criterion for bioequivalence analysis was that the 90% confidence interval for the Test/Reference ratio of AUC0-∞ geometric means was within the 80.00-125.00 range; p < 0.0001, ANOVA; Geometric Mean Ratio = 111.83, 90% CI 2-sided [108.19 to 115.29]

5. Secondary Outcome: Description Tmax: Time to Achieve Cmax Reference
Description: The results will be displayed and summarised in tables and figures.
Time Frame: 0 h (pre-dose), 15, 30, 45 min, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24 and 36 h after drug administration
Measure: Median (Full Range); unit: h
Groups:
- Riluzole Orodispersible Film (Test): The subjects will be treated with one orodispersible film containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence.
  The subjects received single oral doses of 50 mg of riluzole, as test orodispersible film , in 2 of 4 subsequent periods separated by wash-out intervals of at least 7 days between consecutive administrations, according to a 2-treatment, 4-period, replicate cross-over design.
Arm/Group | Riluzole Orodispersible Film (Test) | Rilutek® Tablet (Reference)
Number analyzed (Participants) | 51 | 51
h | 0.75 [0.25 to 2] | 0.75 [0.25 to 4]

6. Secondary Outcome: Evaluation of the Test Product Palatability
Description: Palatability was scored according to the following scale. Palatability evaluation description and scores (between brackets): Very unpleasant (0), Unpleasant (1), Acceptable (2), Good (3), Very good (4).
  Minimun value is 0, maximum value is 4. An higher score mean a better outcome.
Time Frame: Immediately after 1st Test product administration, approximately within 5 minutes after administration
Population: Data for this outcome measure were only collected after administration of the Test product (Riluzole orodispersible film). The overall number of participants analyzed is the number of subjects who received Riluzole 50 mg orodispersible film (T) at the 1st administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Riluzole Orodispersible Film (Test)
Number analyzed (Participants) | 52
Participants
  0 - very unpleasant | 0
  1 - unpleasant | 1
  2 - acceptable | 15
  3 - good | 31
  4 - very good | 5

7. Secondary Outcome: Evaluation of the Test Product Palatability
Description: as for outcome 6
Time Frame: Immediately after 2nd Test product administration, approximately within 5 minutes after administration
Population: Data for this outcome measure were only collected after administration of the Test product (Riluzole orodispersible film). The overall number of participants analyzed is the number of subjects who received Riluzole 50 mg orodispersible film (T) at the 2nd administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Riluzole Orodispersible Film (Test)
Number analyzed (Participants) | 51
Participants
  0 - very unpleasant | 0
  1 - unpleasant | 2
  2 - acceptable | 14
  3 - good | 28
  4 - very good | 7

8. Secondary Outcome: Number of Participants With Mucosal Irritation
Description: Mouth inspections were performed before the Test administration and 30 min and 1 h after administrations of Test, to check the mucosal irritation at the application site. The outcome number shows the overall number of subjects with mucosal irritation.
Time Frame: pre-dose (0), 0.5 and 1 h after the drug administration
Population: Data for this outcome measure were only collected for the Test product (Riluzole orodispersible film). No mouth inspection was performed after Reference (Rilutek®) administration. The overall number of participants analyzed is the number of subjects who received Riluzole 50 mg orodispersible film (T).
Measure: Count of Participants; unit: Participants
Arm/Group | Riluzole Orodispersible Film (Test)
Number analyzed (Participants) | 52
Participants | 0

9. Secondary Outcome: Haematology, Blood Chemistry and Urinalysis Laboratory Tests Interpretation
Description: Overall investigator's interpretation (as normal or abnormal and, if abnormal, clinically significant or not clinically significant).
  The following analyses were performed at screening: Leukocytes, erythrocytes, haemoglobin, haematocrit, MCV, MCH, MCHC, thrombocytes, electrolytes, enzymes (alkaline phosphatase, γ-GT, AST, ALT), total bilirubin, creatinine, glucose, urea, uric acid, total cholesterol, triglycerides, cotinine, total proteins. Serum pregnancy test (women). Urine analysis: pH, specific weight, appearance, colour, nitrites, proteins, glucose, urobilinogen, bilirubin, ketones, haematic pigments, leukocytes. Urine sediment (analysis performed only if positive): leukocytes, erythrocytes, flat cells, round cells, crystals, cylinders, mucus, bacteria. Hepatitis B (HBs antigen), Hepatitis C (HCV antibodies), HIV 1/2 (HIV Ag/Ab combo).
  The same analyses, with the exception of cotinine, urine drug test, virology and pregnancy test, were performed at the final visit
Time Frame: At screening (initial visit) and at final visit (approximately 1 month)
Measure: Count of Participants; unit: Participants
Groups:
- Riluzole Orodispersible Film (Test) / Rilutek® Tablet (Reference): The evaluation of the laboratory parameters was carried out at screening and final visit, without a partition of treatment group.
Arm/Group | Riluzole Orodispersible Film (Test) / Rilutek® Tablet (Reference)
Number analyzed (Participants) | 53
Participants
  Screening visit: Normal | 3
  Screening visit: Abnormal, Not Clinically Significant | 50
  Screening visit: Abnormal, Clinically Significant | 0
  Final visit (approximately 1 month): Normal | 1
  Final visit (approximately 1 month): Abnormal, Not Clinically Significant | 52
  Final visit (approximately 1 month): Abnormal, Clinically Significant | 0

ADVERSE EVENTS:
Time Frame: 36 days
Groups:
- Rilutek® (Reference): The subjects were treated with one film-coated table containing 50 mg of riluzole in two out of the four study periods according to the randomisation sequence
  Rilutek 50Mg Tablet: One film-coated tablet was swallowed (without chewing) with 150 mL of still mineral water.
Arm/Group | Riluzole Orodispersible Film (Test) | Rilutek® (Reference)
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/53
Other Adverse Events (participants affected / at risk) | 52/52 | 14/53
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riluzole Orodispersible Film (Test) (N=52) | Rilutek® (Reference) (N=53)
Hypoaesthesia oral (Gastrointestinal disorders) | 52 (102) | 0 (0)
Headache (Nervous system disorders) | 11 (15) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT04819438/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-31): https://cdn.clinicaltrials.gov/large-docs/38/NCT04819438/SAP_001.pdf